CLINICAL TRIAL: NCT02997514
Title: Implementation and Evaluation of Solution Focused Coaching Strategy Within a Paediatric Multidisciplinary Neuromuscular Clinic
Brief Title: Solution Focused Coaching Strategy Within a Paediatric Multidisciplinary Neuromuscular Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: AHSC AFP Innovation Fund- Ontario Government (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-651
Record Dates: First submitted 2016-11-30; First posted 2016-12-20 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2018-07

CONDITIONS: Neuromuscular Diseases
Keywords: Solution focused coaching; Self determination
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Solution Focused Coaching (Active Comparator): Participants will engage in 5 solution focused coaching sessions, each up to 60 minutes in duration
  Interventions: Behavioral: Intensive Solution Focused Coaching
- Solution Focused Coaching (Active Comparator): Participants will engage in 1 solution focused coaching session up to 60 minutes in duration
  Interventions: Behavioral: Solution Focused Coaching

INTERVENTIONS:
Behavioral: Solution Focused Coaching — SFC is an approach that uses strategic questioning to help the client envision what they would like to be different and how they will take action towards achieving their goals.
  Arms: Solution Focused Coaching
Behavioral: Intensive Solution Focused Coaching — Intensive SFC is an approach that uses strategic questioning to help the client envision what they would like to be different and how they will take action towards achieving their goals.
  Arms: Intensive Solution Focused Coaching

SUMMARY:
The purpose of this study is to implement Solution Focused Coaching in pediatric rehabilitation (SFC-peds) within the multidisciplinary neuromuscular clinic at Holland Bloorview Kids Rehabilitation Hospital and evaluate its effect on children's ability to set and attain personally meaningful goals. A secondary goal is to determine the impact of SFC-peds on self-determination in children with neuromuscular conditions. This study aims to compare two methods of SCF-peds delivery, a single coaching session vs. intensive coaching (5 sessions) on goal attainment. This study will also help researchers and clinicians understand the types of goals that are set by children with neuromuscular conditions. Lastly, this study is going to explore with the participants their perception of the feasibility of using this methodology within a clinical context.

DETAILED DESCRIPTION:
Nationally, standards of care have been published for paediatric neuromuscular (NM) conditions to optimize care, improve quality of life and increase life span. Children with NM conditions are followed in regional multidisciplinary clinics in Ontario and across Canada. At each visit they can be seen by 8 health care providers each focusing on and making recommendations for the different aspects of their care. Currently, there are no evidenced based interventions for children with NM conditions evaluating the ability of children to set and attain their care goals and/or other personally meaningful goals.

Self-determination is defined as the ability to "use skills, knowledge and beliefs that enable a person to engage in goal directed, self-regulated, autonomous behavior." The development of self-determination is a process that begins in childhood. Solution Focused Coaching (SFC) is a strengths- based, client-centered approach to service delivery that supports clients to build on their existing capacity to move closer to meaningful goals. This study will evaluate the impact of SFC on goal setting, achievement and self determination in children with NM conditions.

ELIGIBILITY:
Inclusion Criteria:

* child has a primary NM diagnosis
* child ages 10-18 years
* child able to converse orally in English
* child has a willingness to engage in the coaching intervention
* child is aware that they have a neuromuscular condition
* child is followed clinically in the Neuromuscular Clinic at Holland Bloorview Kids Rehabilitation Hospital at 4-6 month intervals
* child has internet access at home and a device to connect to the internet with a camera
* child is able to demonstrate capacity to consent
* parent is able to read and write in English

Exclusion Criteria:

-child has a moderate to severe intellectual disability

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Change on Canadian Occupational Performance Measure (COPM) | Week 0 and Week 14
Change on Goal Attainment Scaling (GAS) | Week 0 and Week 14

SECONDARY OUTCOMES:
American Research Council's Self Determination Scale (ARC SDS) | Week 0 and Week 14
Solution-Focused Fidelity Instrument (SFFI) | Weeks: 2, 3, 4, 6, 10 and 14
  Done after each coaching session
Thematic Analysis of Interview Questions Exploring Solution Focused Coaching Process | Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Laura McAdam, MD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baldwin P, King G, Evans J, McDougall S, Tucker MA, Servais M. Solution-focused coaching in pediatric rehabilitation: an integrated model for practice. Phys Occup Ther Pediatr. 2013 Nov;33(4):467-83. doi: 10.3109/01942638.2013.784718. Epub 2013 Apr 24. PMID 23611310
- [Background] Field, S., Martin, J., Miller, R., Ward, M., & Wehmeyer, M. (1998). A practical guide for teaching self-determination. Reston, VA: Council for Exceptional Children. In Field, S., Martin, J., Miller, R., Ward, M., & Wehmeyer, M. (1998). Self-determination for persons with disabilities: A position statement of me division on career development and transition. Career Development for Exceptional Individuals, 21(2), 113-128.